CLINICAL TRIAL: NCT03338842
Title: Virtual Reality Treatment for Phantom Limb Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Moss Rehabilitation Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 823287
Record Dates: First submitted 2017-11-01; First posted 2017-11-09 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Lower Limb Amputation Above Knee (Injury); Lower Limb Amputation Below Knee (Injury); Phantom Limb Pain
MeSH Terms: conditions — Wounds and Injuries; Phantom Limb

STUDY DESIGN:
Intervention Model Description: In the first phase (A), subjects will receive the Distraction VR treatment during 5, 6, or 7 one-hour-long sessions occurring twice weekly. After the A phase, the remaining sessions (B phase) will consist of Lower-Limb VR treatment. This number includes a mean of 6 (range 5-7) phase A sessions and mean of 11 (range 10-12) phase B sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Distractor and Lower limb VR (Experimental): The training sessions consist of Phase 1 (Distractor VR) in which patients will explore VR environments and Phase 2 (Lower limb VR) in which they will play games using their VR lower-limbs.
  Interventions: Device: Distractor and Lower limb VR

INTERVENTIONS:
Device: Distractor and Lower limb VR — In the first phase (A), subjects will receive the Distraction VR treatment during 5, 6, or 7 one-hour-long sessions occurring twice weekly. After the A phase, the remaining sessions (B phase) will consist of Lower-Limb VR treatment. This number includes a mean of 6 (range 5-7) phase A sessions and mean of 11 (range 10-12) phase B sessions.

SUMMARY:
Patients with limb amputations experience the sensation of the missing extremity, which is sometimes coupled with a persistent and debilitating pain in the missing limb, a condition known as phantom limb pain (PLP). This study will test the use of virtual reality (VR) training as a possible treatment of PLP.

DETAILED DESCRIPTION:
Approximately 90% of patients with limb amputations experience the persistent sensation of the missing extremity, a phenomenon known as phantom limb (PL). Most patients with PL also experience a persistent and debilitating pain in the missing limb, a condition known as phantom limb pain (PLP).PLP is often attributed to a disruption of the primary sensory-motor representation, generating "noise" in the representation of the missing extremity, manifesting as pain. If loss of sensory feedback causes degradation of the these cortices, interventions that provide visual feedback about the missing extremity might fine-tune the primary sensory-motor cortices, thereby reducing pain. Within this framework, the present study explores the use of virtual reality (VR) training as a possible treatment of PLP. Twenty-five subjects with lower-limb amputation and chronic PLP will undergo a Virtual Reality (VR) treatment (17 one-hour sessions) consisting in two phases: a Distraction VR phase (5-7 sessions) in which they will explore VR environments using a joystick and a Lower-Limb VR treatment phase (10-12 sessions) in which they will participate in a variety of games and activities using their VR lower-limbs. A comprehensive battery for the assessment of the characteristics, intensity and the daily-life implication of PLP will be presented before and after the treatment and in three follow up testing sessions (1,4, 8 weeks). Furthermore, pain intensity will be assessed before and after each VR session. A dramatic reduction of PLP is expected after the VR treatment and that these beneficial effects remain stable in time.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will have undergone amputation of one leg (either above or below the knee) at least 4 months before the enrollment in the study;
* Will have chronic pain in the phantom limb:

Exclusion Criteria:

* History of stroke or traumatic brain injury;
* Major active psychiatric illness that may interfere with required study procedures or treatments as determined by the PI on the study, who is a behavioral neurologist;
* Subjects with major medical illness that would be expected to interfere with their ability to complete the study will be excluded.
* Subjects with implanted electronic devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Changes in the Brief Pain Inventory | Pre and post Phase 1; Pre and post Phase 2; at 1, 4 and 8 weeks
  The Brief Pain Inventory is a questionnaire which provide a description of the type and location of pain (question 1-2),the pain severity (question 3-6 pain rating scales with 0-10 range - with 10 indicating severe pain), of the current treatment for pain (question 7-8) and the pain interference in daily life (question 9- range from 0 to 10 with a maximum score of 10 indicating severe interference). A decrease (i.e. reduction in the scores) in pain severity and in the pain interference in daily activity is expected as consequence of the virtual reality training.
Changes in the McGill Pain Questionnaire | Pre and post Phase 1; Pre and post Phase 2; at 1, 4 and 8 weeks
  The McGill Pain Questionnaire is a questionnaire which provide a description of the type of pain using series of adjectives on of the pain severity, using a visual analogue scale (range of 0-100 range - with 100 indicating severe pain). A decrease in pain severity (decrease in the score in the visual analogue scale) is expected as consequence of the virtual reality training.
Changes in the Frenchay Activities Index | Pre and post Phase 1; Pre and post Phase 2; at 1, 4 and 8 weeks
  The the Frenchay Activities Index is a 15 items questionnaire, which investigate how often people perform certain daily activity (e.g. preparing meals), using a scale from 0 to 3, with a score of 3 indicating that the activity is performed frequently. An increase in the Frenchay Activities Index is expected as consequence of the virtual reality training.
Changes in the12-Item Short Form Health Survey | Pre and post Phase 1; Pre and post Phase 2; at 1, 4 and 8 weeks
  The12-Item Short Form Health Survey is a questionnaire which investigate the quality of emotional and physical heath of individuals. An improvement in the quality of the individuals' health is expected as consequence of the training.
Changes in the Hospital Anxiety and Depression Scale | Pre and post Phase 1; Pre and post Phase 2; at 1, 4 and 8 weeks
  The Hospital Anxiety and Depression Scale measures depression is a 14 questions scale, which measure the level of depression and anxiety (maximum score of 21 indicating abnormal performance). A decrease in the score in this scale is expected as consequence of the virtual reality training

SECONDARY OUTCOMES:
Changes in the Limb deficiency and Phantom Limb questionnaire. | Pre and post Phase 1; Pre and post Phase 2; at 1, 4 and 8 weeks
  The Limb Deficiency and Phantom Limb questionnaire investigate qualitatively the phantom limb sensations.A reduction in the reported phantom limb sensation is expected as consequence of the virtual reality training
Changes in the 13-item Pain Catastrophizing scale | Pre and post Phase 1; Pre and post Phase 2; at 1, 4 and 8 weeks
  The 13-item Pain Catastrophizing scale assesses the level of negative thoughts and feeling associated with pain using a scale from 0-4 (score of 4 indicating highest frequency; maximum overall score 52). A reduction of the overall score is expected after the virtual reality training

CONTACTS AND LOCATIONS:
Overall Officials: Branch Coslett, Principal Investigator — hbc@mail.med.upenn.edu; Laurel Buxbaum, Principal Investigator — Lbuxbaum@einstein.edu
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weeks SR, Anderson-Barnes VC, Tsao JW. Phantom limb pain: theories and therapies. Neurologist. 2010 Sep;16(5):277-86. doi: 10.1097/NRL.0b013e3181edf128. PMID 20827116
- [Background] Dietrich C, Walter-Walsh K, Preissler S, Hofmann GO, Witte OW, Miltner WH, Weiss T. Sensory feedback prosthesis reduces phantom limb pain: proof of a principle. Neurosci Lett. 2012 Jan 24;507(2):97-100. doi: 10.1016/j.neulet.2011.10.068. Epub 2011 Nov 7. PMID 22085692
- [Background] Chan BL, Witt R, Charrow AP, Magee A, Howard R, Pasquina PF, Heilman KM, Tsao JW. Mirror therapy for phantom limb pain. N Engl J Med. 2007 Nov 22;357(21):2206-7. doi: 10.1056/NEJMc071927. No abstract available. PMID 18032777
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Melzack R. The short-form McGill Pain Questionnaire. Pain. 1987 Aug;30(2):191-197. doi: 10.1016/0304-3959(87)91074-8. PMID 3670870
- [Background] Holbrook M, Skilbeck CE. An activities index for use with stroke patients. Age Ageing. 1983 May;12(2):166-70. doi: 10.1093/ageing/12.2.166. PMID 6869117
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Goller AI, Richards K, Novak S, Ward J. Mirror-touch synaesthesia in the phantom limbs of amputees. Cortex. 2013 Jan;49(1):243-51. doi: 10.1016/j.cortex.2011.05.002. Epub 2011 Jun 22. PMID 22981809